CLINICAL TRIAL: NCT06933251
Title: Clinical Study of PCSK9 Inhibitor and PD-1 Inhibitor Combined With Neoadjuvant Chemoradiotherapy in the Treatment of pMMR/MSS Locally Advanced Rectal Cancer
Brief Title: PCSK9 Inhibitor and PD-1 Inhibitor Combined With Neoadjuvant Chemoradiotherapy for pMMR/MSS Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lron-Man 03
Record Dates: First submitted 2025-03-06; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: neoadjuvant chemoradiotherapy; PD-1 inhibitor; PCSK9 inhibitor; pMMR/MSS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Chemoradiotherapy Combined with Immunotherapy and PCSK9 inhibitor Treatment (Experimental): Building on short-term radiotherapy combined with chemotherapy, the treatment integrates PD-1 inhibitor immunotherapy and PCSK9 inhibitor therapy.
  Interventions: Drug: Neoadjuvant Chemoradiotherapy Combined with PD-1 inhibitor Immunotherapy and PCSK9 Inhibitor Therapy

INTERVENTIONS:
Drug: Neoadjuvant Chemoradiotherapy Combined with PD-1 inhibitor Immunotherapy and PCSK9 Inhibitor Therapy — 1. Neoadjuvant Treatment 1.1 Short-Course Radiotherapy (SCRT) Total Dose: 25 Gy in 5 fractions over 5 days. Interval: 1-week rest before the next stage. 1.2 Chemotherapy and Immunotherapy Regimen: Start 1 week after SCRT with 6 cycles of CAPOX chemotherapy combined with PD-1 inhibitor immunotherapy (3 weeks per cycle).
     1.3 PCSK9 Inhibitor Administration: Subcutaneous injection every 4 weeks during neoadjuvant therapy (6 cycles total).
  2. Multidisciplinary Team (MDT) Discussion Timing: 2 weeks after completing neoadjuvant therapy.
  Approach:
  Patients achieving clinical complete response (cCR): "Watch-and-wait" strategy. Others: Surgery based on MDT evaluation.

SUMMARY:
This is a single-center, open-label, single-arm clinical study aimed at conducting a preliminary evaluation of the efficacy and safety of combining PCSK9 inhibitors and PD-1 inhibitors (dual inhibitors) with neoadjuvant chemoradiotherapy in patients with pMMR/MSS locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study aims to evaluate the complete response (CR) rate of PCSK9 inhibitor and PD-1 inhibitor combination therapy (dual inhibitors) in conjunction with neoadjuvant chemoradiotherapy for patients with pMMR/MSS locally advanced rectal cancer. Specifically, the study will assess the pathological complete response (pCR) rate two weeks after neoadjuvant therapy, the clinical complete response (cCR) rate under the "watch-and-wait" strategy, objective response rate (ORR), R0 resection rate, tumor regression grade (TRG), and sphincter preservation rate. Additionally, the study will evaluate the 2-year disease-free survival (DFS) and overall survival (OS) following dual-inhibitor combined neoadjuvant chemoradiotherapy. The safety and tolerability of this combination therapy will also be comprehensively assessed based on NCI-CTCAE 4.03 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, regardless of gender;
2. Histologically confirmed pMMR/MSS rectal adenocarcinoma, with clinical staging of cT3/T4 or cN+, and tumor located ≤12 cm from the anal verge;
3. No distant metastasis;
4. ECOG performance status of 0-1;
5. Baseline hematological and biochemical parameters meet the following criteria: neutrophils ≥1.5×10^9/L, hemoglobin ≥90 g/L, platelets ≥100×10^9/L, ALT/AST ≤2.5 ULN, creatinine ≤1 ULN;
6. Good compliance and willingness to sign an informed consent form.

Exclusion Criteria:

1. History of allergies to PCSK9 monoclonal antibody, PD-1 monoclonal antibody, capecitabine, or oxaliplatin;
2. Preoperative pathological diagnosis of non-pMMR/MSS rectal adenocarcinoma;
3. Use of other long-term lipid-lowering drugs leading to conditions such as hypolipidemia;
4. Pregnant or breastfeeding women;
5. History of other malignancies within the past 5 years;
6. Previous history of anti-tumor treatments, including radiotherapy, chemotherapy, immune checkpoint inhibitors, T-cell related therapies, etc.;
7. History of severe neurological or psychiatric disorders (e.g., schizophrenia, dementia, or epilepsy);
8. Current severe cardiovascular disease (heart failure or arrhythmia), renal insufficiency, or liver dysfunction; Note: Whether the patient can tolerate the specific treatment or measures should be assessed by a cardiologist based on the patient's condition.
9. Acute myocardial infarction or ischemic stroke within 6 months prior to enrollment;
10. Presence of uncontrolled infections requiring systemic treatment;
11. Active autoimmune diseases or immunodeficiencies, a history of organ transplantation, or systemic use of immunosuppressive agents;
12. Known history of HIV infection (e.g., HIV 1-2 antibody positive), active syphilis, or active pulmonary tuberculosis;
13. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection during screening (e.g., HBsAg positive, HBV DNA positive, HCV RNA positive, or anti-HCV antibody positive);
14. Known allergy to any component of the treatment;
15. Investigator's judgment that other factors exist which may cause early termination of the trial, such as severe disease (including psychiatric disorders), alcohol abuse, drug use, or social or familial factors affecting patient safety or compliance;
16. History of hypocholesterolemia (total cholesterol [TC] <3.6 mmol/L or <140 mg/dL, low-density lipoprotein cholesterol [LDL-C] <1.8 mmol/L or <70 mg/dL, high-density lipoprotein cholesterol [HDL-C] <1.0 mmol/L [male] or <1.3 mmol/L [female]), hypolipidemia (triglycerides [TG] <0.5 mmol/L or <45 mg/dL), or a family history of these conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
CR | pCR :within 2 weeks after surgery; cCR :2 weeks after radiotherapy ends
  complete response rate=(number of pathological complete responses + number of clinical complete responses)/total number of patients
AE rate | During neoadjuvant chemoradiotherapy combined with immunotherapy, an average of 6 months
  Adverse event rate

SECONDARY OUTCOMES:
DFS | 5 years
  Disease-free survival
OS | 5 years
  Overall survival time
ORR | within 2 weeks after surgery
  objective response rate
TRG | At the time of postoperative pathological assessment (within 1 week after surgery)
  Tumor regression grade
OPR | immediately after surgery
  organ preservation rate

CONTACTS AND LOCATIONS:
Locations (1):
- No. 106, Zhongshan 2nd Road, Yuexiu District, Guangzhou, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Bao X, Hu M, Chang H, Jiao M, Cheng J, Xie L, Huang Q, Li F, Li CY. Inhibition of PCSK9 potentiates immune checkpoint therapy for cancer. Nature. 2020 Dec;588(7839):693-698. doi: 10.1038/s41586-020-2911-7. Epub 2020 Nov 11. PMID 33177715
- [Background] Yuan J, Cai T, Zheng X, Ren Y, Qi J, Lu X, Chen H, Lin H, Chen Z, Liu M, He S, Chen Q, Feng S, Wu Y, Zhang Z, Ding Y, Yang W. Potentiating CD8+ T cell antitumor activity by inhibiting PCSK9 to promote LDLR-mediated TCR recycling and signaling. Protein Cell. 2021 Apr;12(4):240-260. doi: 10.1007/s13238-021-00821-2. Epub 2021 Feb 19. PMID 33606190